CLINICAL TRIAL: NCT05785364
Title: Monocer Cup: Open, Prospective, Multicentric, Non Randomised Observational Study
Brief Title: A Post Market Surveillance Study About the MONOCER Cup
Status: Recruiting | Type: Observational
Sponsor: Medacta International SA (Industry)
Responsible Party: Sponsor
Other Study IDs: P01.026.02
Record Dates: First submitted 2023-03-13; First posted 2023-03-27 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Total Hip Arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Mpact 3D metal MONOCER cup — adult patients requiring a total hip arthroplasty under 75 years old, will receive the Mpact 3D metal cup, as acetabular sheel device implanted

SUMMARY:
Over the years, the use of large diameter femoral heads has become increasingly common in orthopaedics due to the decreased risk of dislocation due to increased jumping distance and range of motion. The history of total hip arthroplasty does not favour large diameter heads, especially as conventional polyethylene has a high risk of wear. The development of hard-on-hard bearings (CoC) with a second generation ceramic material and the introduction of cross-linked PE have led to the reintroduction of this concept. The Mpact 3D Metal MonoCER cup was developed to offer the advantages of accommodating large diameter heads with an external metal cup with a pre-assembled system that avoids the surgical step of insert-cotile coupling.

DETAILED DESCRIPTION:
All patients candidated to receive a total hip arthroplasty under 75 years old, who will receive a Mpact 3D Metal cup will be proposed to take part to the study. They will receive the same treatment in case they will not partecipate; the study is an observational study according to standard practice. The study aim to assess the long term peformance of the cup at 10 years after surgery. The patients will be visited at 6 months, 1, 5 and 10 years after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing total hip arthroplasty who will receive the Mpact 3D Metal MonoCER acetabular component according to the instructions for use
2. Patients who have signed the informed consent to participate in the study

Exclusion Criteria:

1. Minor patients, patients over 75 years of age at the time of primary surgery;
2. Any patient who is unable or unwilling to give informed consent to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients listed for a Total Hip Arthroplasty (THA) with Mpact 3D Metal MONOCER cup, meeting all inclusion/exclusion criteria, at the research site, will be proposed to take part to the current study during the preoperative visit.
  The investigator will explain to each participant the nature of the study, its purpose, the procedures involved, the expected duration, the potential risks and benefits and any discomfort it may entail
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-01-25 (Actual); Primary Completion 2050-02-01 (Estimated); Study Completion 2050-02-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of implant survivorship using Kaplan Meier curve | 10 years
  a Kaplan Meir survival curve will be calcuated

SECONDARY OUTCOMES:
Assessment of Device stability throught a radiological exam | 6 months, 1 year, 5 and 10 years
  standard x-ray examination will be peformed during the visits
Assessment of the clinical outcome following total hip replacement using the Harris Hip score | 6 months, 1 year, 5 and 10 years
  HHS score will be completed
Device Safety assessed through adverse event collection | up to 10 yrs follow-up
  number of adverse event occurred

CONTACTS AND LOCATIONS:
Overall Officials: Placido Bartolone, Dr, Principal Investigator — Hirslanden, Clinique la Colline 76A Av. de la Roseraie 1205 Genève
Locations (1):
- Hirslanden, Clinique la Colline, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No